CLINICAL TRIAL: NCT02007278
Title: Glycemic Excursions in Type 2 Diabetic Patients Treated With Vildagliptin and Metformin (GalvusMet) Versus Glimepiride and Metformin
Brief Title: Glycemic Excursions in Type 2 Diabetic Patients With Vildagliptin and Metformin Versus Vildagliptin and Glimepiride
Acronym: GLOBE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ACO01
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes; Hypoglycemia
Keywords: diabetes; hypoglycemia; glycemic variability; vildagliptin; glimepiride
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Diabetes Mellitus | interventions — Vildagliptin; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vildagliptin and metformin (Active Comparator): Based on basal dose of metformin, administration of vildagliptin/metformin 50 mg/850 mg twice daily (bid) or 50 mg/1000 mg bid for 12 weeks
  Interventions: Drug: vildagliptin and metformin (combination)
- glimepiride and metformin (Active Comparator): Protocol specified dosage and frequency of glimepiride + metformin for 12 weeks based on basal dose of metformin
  Interventions: Drug: glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: vildagliptin and metformin (combination) — vildagliptin and metformin combination therapy as 50mg/850mg bid or 50mg/1000mg bid
  Arms: vildagliptin and metformin
Drug: glimepiride
  Arms: glimepiride and metformin
Drug: Metformin
  Arms: glimepiride and metformin

SUMMARY:
The purpose of this study was to compare the effect of a fixed dose combination of vildagliptin plus metformin versus combination therapy of glimepiride plus metformin in glycemic variability in patients with type 2 diabetes who have not achieved adequate control of their disease prior to treatment with metformin monotherapy in optimal doses.

ELIGIBILITY:
Key Inclusion Criteria:

* HbA1c between 8%-10.5% in stable metformin dose (>1500 mg/day), four weeks prior visit 1

Key Exclusion Criteria:

* Use of other antidiabetic oral therapy during the last 3 months (sulphonylurea, glitazones, GLP-1 analogues, DPP-4 inhibitors), except metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Colombia (8):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Manizales, Caldas Department
  - Novartis Investigative Site, Cali, Colombia
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Chía, Cundinamarca
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Montería

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9 research centers participated in the study, from which 76 patients were screened for inclusion and exclusion criteria, obtaining 40 patients eligible for randomization
Period: Overall Study
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Started | 20 | 20
Completed | 18 | 17
Not Completed | 2 | 3
Not completed — Failure to comply with an eligibility | 0 | 1
Not completed — Ingestion of drugs not allowed in study | 0 | 1
Not completed — Incorrect medication administration | 1 | 0
Not completed — Mis-randomization | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set
Groups:
- Total: Total of all reporting groups
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.74 (10.58) | 55.70 (11.51) | 56.25 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Variability Measured by Mean Amplitude of Glucose Excursions (MAGE)
Description: Mean Amplitude of Glycemic Excursions (MAGE) , which determines the average blood glucose excursions either above or below a value of one standard deviation of the average value of glucose in a given day. MAGE is calculated from the data of continuous tissue glucose monitoring obtained during the measurement period. MAGE is calculated with the formula Σ λ / χ if λ> ν (where λ = changes in blood glucose from peak to nadir, χ = number of valid observations, ν = 1 standard deviation of the mean glucose during a period of 24 hours) from the data of continuous monitoring of the tissue glucose, obtained during the period of measurement.
Time Frame: Week 12
Population: Analysis set includes all randomized patients excluding the ones who were prematurely withdrawn and the ones who have no data from visit 7 which required for comparison.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 16 | 16
mg/dL | 6.68 (1.48) | 6.23 (1.08)
Statistical Analysis 1: Comparison: Vildagliptin and Metformin vs Glimepiride and Metformin; Test type: Non-Inferiority or Equivalence — Power=95%; significance level=5%, characteristic operation curves were used with a non-central F distribution for the calculation of the sample size; p = 0.4510, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Glycemic Variability Measured by Continuous Overlapping Net Glycemic Action (CONGA)
Description: Continuous Overlapping Net Glycemic Action (CONGA) which assesses intra-day glycemic variability by calculating the difference between values at different intervals, adjusted according to requirements with the advantage of being highly reproducible.
  CONGA is calculated in the conventional way with the formula √tқΣt = t1 (Dt -Ď2) / қ - 1, Ď = tқ Σ Dt t = t1 / қ, Dt = Gt-Gt-m (where қ = Observations with an observation n x 60 minutes, G = glucose measure) from the data of continuous monitoring of tissue glucose obtained during the measurement period.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 16 | 16
mg/dL | 2.92 (0.93) | 3.01 (1.10)

3. Secondary Outcome: Glycemic Variability Measured by Total Standard Deviation (TSD)
Description: Total standard deviation (TSD) or standard deviation of all values of a given measurement period, which has the advantage of being able to include all measured values on a given time period (even several days) through a common and simple statistical concept.
  TSD is calculated conventionally with the formula σ = √Σ (Xi - ῦ) 2 / N (where Xi represents each of the values, ῦ represents the population mean and N is the number of observations) from the data of continuous monitoring of tissue glucose obtained during the measurement.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 16 | 16
mg/dL | 1.36 (0.40) | 1.40 (0.42)

4. Secondary Outcome: Percentage of Patients Who Achieved a Decrease Equal to or Greater Than 0.3% in Value of HbA1c at Week 12
Time Frame: Screening visit , 12 weeks of treatment
Population: Analysis set includes all randomized patients excluding the ones who were prematurely withdrawn and the ones who have confirmed non-concordant data
Measure: Number; unit: percentage of patients
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 17 | 17
percentage of patients | 100.0 | 100.0

5. Secondary Outcome: Change in HbA1c at Week 12 of Treatment in Comparison to HbA1c at Baseline
Time Frame: baseline, 12 weeks of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 17 | 17
Percentage of glycosylated haemoglobin | 1.92 (1.1) | 2.28 (0.79)

6. Secondary Outcome: Number of Patients With Incidence of Hypoglycemia
Description: Hypoglycemia defined as Glycemia < 70 mg/dl
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 16 | 16
Patients | 1 | 4

7. Secondary Outcome: Mean Amplitude of Glycemic Excursions (MAGE) for Patients With Hypoglycemia Incidence After 12 Weeks of Treatment
Description: MAGE , which determines the average blood glucose excursions either above or below a value of one standard deviation of the average value of glucose in a given day. MAGE is calculated from the data of continuous tissue glucose monitoring obtained during the measurement period. MAGE is calculated with the formula Σ λ / χ if λ> ν (where λ = changes in blood glucose from peak to nadir, χ = number of valid observations, ν = 1 standard deviation of the mean glucose during a period of 24 hours) from the data of continuous monitoring of the tissue glucose, obtained during the period of measurement. In this endpoint, mean MAGE value is reported for hypo glycemic patients.
Time Frame: 12 weeks
Population: Analysis set includes all randomized patients excluding the ones who were prematurely withdrawn and the ones who have no data from visit 7 which required for comparison and had at least one hypoglycemia event.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 1 | 4
mg/dL | 5.23 (NA) — Standard deviation is not measurable for one patient | 5.53 (0.82)

8. Secondary Outcome: Number of Patients With Any Adverse Events, Serious Adverse Events and Death
Time Frame: 12 weeks
Population: All the randomized patients.
Measure: Number; unit: Patients
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Number analyzed (Participants) | 20 | 20
Patients
  Any adverse events (serious and non-serious) | 9 | 13
  Serious Adverse Events | 0 | 1
  Death | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vildagliptin and Metformin | Glimepiride and Metformin
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 9/20 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin and Metformin (N=20) | Glimepiride and Metformin (N=20)
Erysipelas (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin and Metformin (N=20) | Glimepiride and Metformin (N=20)
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 1
Presbyopia (Eye disorders) | 0 | 1
Refraction disorder (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Hypothermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 3 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Chikungunya virus infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 3
Urine abnormality (Renal and urinary disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.